CLINICAL TRIAL: NCT02521480
Title: Determination of the Analgesic Effects of One Session of Postoperative Left Prefrontal Cortex Repetitive Transcranial Magnetic Stimulation (TMS) Following Vaginal Reconstructive Surgery.
Brief Title: Determination of Analgesic Effect From One Transcranial Magnetic Stimulation(TMS)Treatment Following Vaginal Reconstructive Surgery.
Acronym: TMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not feasible or convenient for the subject
Sponsor: East Tennessee State University (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Principal Investigator, Dr. Norman Moore, Norman Moore, M.D., East Tennessee State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0615.11f
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Transcranial Magnetic Stimulation (Active Comparator): During TMS treatment, a coil, which creates a magnetic field, will be placed on the left prefrontal area of the head. Active TMS will stimulate for 4 seconds, pause for 26 seconds, and repeat this for approximately 40 minutes. There will be a total of 3000 pulses during treatment. We expect TMS to decrease pain and depression.
  Interventions: Device: Active Transcranial Magnetic Stimulation
- Sham Transcranial Magnetic Stimulation (Sham Comparator): During sham TMS, a coil will be placed on the left prefrontal area of the head. Sham TMS will simulate active treatment as described in active arm.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active Transcranial Magnetic Stimulation — TMS is a non-invasive treatment. During TMS treatment, a coil, which creates a magnetic field, will be placed on the left prefrontal area of the head. Active TMS will stimulate for 4 seconds, pause for 26 seconds, and repeat this for approximately 40 minutes. There will be a total of 3000 pulses during treatment. We expect TMS to decrease pain and depression. In order to find out if this is true, we will compare real TMS with sham (inactive) TMS.This will allow us to decide if active TMS is successful because of electrical stimulation, or because of the support, concern, and understanding of the research team.
  Arms: Active Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Inactive treatment (simulation of active TMS)
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
To determine whether real TMS is more effective than sham TMS in reducing pain following surgery

DETAILED DESCRIPTION:
To determine the amount of opiate and pain medication administered in the week following surgery. Subjects will receive an identical pain control regimen. Participants will undergo TMS motor threshold assessment at the ETSU Innovation Lab prior to the planned surgery. At this appointment a baseline Beck Depression Inventory (BDI), Center for Epidemiological Studies 10-item Depression scale (CES-D) and visual analog scale (VAS) ratings of pain and mood will be obtained.VAS ratings will also be done each evening over the following week. One day after surgery, the subject will return to the Innovation lab for TMS. A total of 22 subjects will be recruited for the study. At the return visit, 11 will receive 40 minutes of 10 Hz repetitive TMS at 120% of rMT (4-second stimulation trains with 26-second interstimulus intervals). The other 11 participants will receive sham treatment under identical settings. Participants, medical staff providing clinical care to patients and raters will not know whether participants receive real or sham TMS. Patients will keep a log of pain medications used over the following week in addition to the VAS ratings. Follow-up will occur one week after the TMS therapy. The subject will turn in logs and repeat BDI and CES-D scales.

ELIGIBILITY:
Inclusion Criteria: Dental fillings, implants, and bridge work are permitted. -

Exclusion Criteria: Metal objects within 30 cm of the brain. These include cochlear implants, stents, vagus nerve stimulators, heart devices, bullet fragments, or jewelry. Monitors, earrings, hearing aids, eyeglasses, jewelry, hair barrettes, cell phones, and digital sound recording device players will be removed. Actively suicidal. Older than 70 years. Seizures, strokes, dementia, or movement disorders. Pregnant or nursing. Permanent makeup with metal ink. Medication known to increase risk of seizures.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Daily and total mg of opiate pain medication and any other over the counter alternate pain medication. | One year

SECONDARY OUTCOMES:
Changes in Visual Analog Scales daily for mood and pain as well as an initial and final Beck Depression Inventory and Center for Epidemiological Studies 10-item Depression Scale | One year

CONTACTS AND LOCATIONS:
Locations (1):
- ETSU Dept. of Psychiatry, Johnson City, Tennessee, United States